CLINICAL TRIAL: NCT04263610
Title: An Open-Label, Randomised, Phase IV Study, to Assess the Efficacy and Safety of Tildrakizumab in Patients With Moderate-to-Severe Chronic Plaque Psoriasis Who Are Non-Responders to Dimethyl Fumarate Therapy (TRANSITION)
Brief Title: Efficacy and Safety of Tildrakizumab in Participants With Moderate-to-Severe Chronic Plaque Psoriasis Who Are Non-Responders to Dimethyl Fumarate Therapy
Acronym: TRANSITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-14745-41; 2019-000817-35 (EudraCT Number)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Plaque Psoriasis
Keywords: Dimethyl fumarate; Tildrakizumab; Moderate-to-severe plaque psoriasis; Chronic Plaque Psoriasis
MeSH Terms: interventions — Dimethyl Fumarate; tildrakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-Germany: Dimethyl fumarate standard scheme (Experimental): Part 1: Participants will receive Dimethyl fumarate (DMF) standard scheme from baseline to Week 16.
  Part 2: Participants achieving a Psoriasis Area and Severity Index (PASI) 75 response (responders) and participants failing to achieve a PASI 75 response but having achieved a PASI 50 response (partial responders) at Week 16 will continue with DMF treatment until Week 40. Participants failing to achieve a PASI 50 response (non-responders) at Week 16 will be treated with Tildrakizumab until Week 40.
  Interventions: Drug: Dimethyl fumarate (DMF) standard scheme; Drug: Tildrakizumab
- Germany: Dimethyl fumarate standard scheme (Experimental): Part 1: Participants will receive DMF standard scheme from Baseline to Week 16. Part 2: Participants achieving a PASI 75 response (responders) and participants failing to achieve a PASI 75 response but having achieved a PASI 50 response (partial responders) at Week 16 will continue with DMF treatment until Week 40. Participants failing to achieve a PASI 50 response (non-responders) at Week 16 will be treated with Tildrakizumab until Week 40.
  Interventions: Drug: Dimethyl fumarate (DMF) standard scheme; Drug: Tildrakizumab
- Germany: Dimethyl fumarate simplified scheme (Experimental): Part 1: Participants will receive DMF simplified scheme from Baseline to Week 16.
  Part 2: Participants achieving a PASI 75 response (responders) and participants failing to achieve a PASI 75 response but having achieved a PASI 50 response (partial responders) at Week 16 will continue with DMF treatment until Week 40. Participants failing to achieve a PASI 50 response (non-responders) at Week 16 will be treated with Tildrakizumab until Week 40.
  Interventions: Drug: Dimethyl fumarate (DMF) simplified scheme; Drug: Tildrakizumab

INTERVENTIONS:
Drug: Dimethyl fumarate (DMF) standard scheme — Participants will receive DMF gastro-resistant tablet orally from baseline to Week 16, at a dose of 30 milligrams (mg) once daily, twice daily, thrice daily in Week 1, Week 2, Week 3 respectively, 120 mg only once in Week 4. Participants will increase DMF dose by 120 mg tablet per week for the subsequent 5 weeks. Participants achieving Psoriasis area and severity Index (PASI) 50-75 (partial responder) or 75 (responder) will continue the DMF treatment until Week 40. The maximum daily dose taken by a participant will be 720 mg.
  Other Names: Skilarence®
  Arms: Germany: Dimethyl fumarate standard scheme; Non-Germany: Dimethyl fumarate standard scheme
Drug: Dimethyl fumarate (DMF) simplified scheme — Participants will receive DMF gastro-resistant tablet orally at a dose of 60, 120, 180, 240, 360 mg daily in Week 1, Week 2, Week 3, Week 4, Week 5 respectively, and 480 mg daily from Week 6 to Week 8. If a PASI is greater than or equal to (>=) 30% at Week 8, no dose increase will be done and if PASI is less than (<) 30% at Week 8, participants will receive 600 mg daily in Week 9 and 720 mg from the Week 10 onwards.
  Other Names: Skilarence®
  Arms: Germany: Dimethyl fumarate simplified scheme
Drug: Tildrakizumab — Participants who achieve PASI less than (<) 50 (non-responders) at Week 16 will receive Tildrakizumab subcutaneous injection at a dose of either 100 or 200 mg [(as per the Summary of Product Characteristics (SmPC)] at Weeks 16, 20 and 32 up to Week 40.
  Other Names: Ilumetri®

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of Tildrakizumab in moderate-to-severe plaque psoriasis participants who are non-responder to Dimethyl fumarate (DMF) at Week 16. The study consists of two parts. Part 1 will include the first 16 weeks of the Treatment Period and Part 2 will include the last 24 weeks of the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written and dated informed consent given before any study related activity is performed
* Participants with at least 6 months history of chronic plaque psoriasis
* Participants diagnosed with moderate-to-severe plaque psoriasis at the Screening Visit
* Candidate for systemic treatment for plaque psoriasis at the Screening Visit

Exclusion Criteria:

* Women currently pregnant, or intend to become pregnant or breastfeeding. Unwillingness/inability for the participants (women or men) to use appropriate measures of contraception (if necessary)
* Other forms of psoriasis than chronic plaque-type
* Participants with drug-induced psoriasis at the Screening Visit
* Participants with history or evidence of skin disease or conditions other than chronic plaque-type psoriasis
* Participants with history of hypersensitivity or allergy to the study drugs
* Concurrent malignancy, current relevant autoimmune diseases other than psoriasis
* Participants with severe renal impairment, haematological abnormality and abnormal liver enzymes at the Screening visit
* Active infectious disease at the Screening Visit
* Participants positive test for human immunodeficiency virus or any other immunosuppressive disease
* Previous exposure to fumarate-based drug or a biologic systemic treatment
* Live vaccination within 4 weeks prior to the Baseline Visit
* Participant who intend to use any concomitant medication with immunomodulating or systemic corticosteroids
* Unable to comply with the requirements of the study or who in the opinion of the study physician should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Part 2: Percentage of Participants Achieving a Psoriasis Area Severity Index 75 (PASI 75) after Tildrakizumab Treatment at Week 40 | Week 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). PASI 75 response, is defined as having an improvement (reduction) of greater than or equal to (>=) 75% in PASI score compared to the baseline score.

SECONDARY OUTCOMES:
Part 1 and Part 2: Percentage of Participants Achieving PASI 50, PASI 75, PASI 90 and PASI 100 (Only for Part 2) Responses | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). PASI 50, 75, 90 response, is defined as having an improvement (reduction) of greater than or equal to (>=) 50%, 75%, 90% and 100% respectively in PASI score compared to the baseline score.
Part 1 and Part 2: Percentage of Participants Achieving an Absolute Psoriasis Area and Severity Index (PASI) Score Less Than or Equal to (<=) 5, 3 and 1 | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Percentage of participants who will achieve an absolute PASI score <= 5, 3 and 1 at Week 8 and Week 16 will be reported.
Part 1 and Part 2: Absolute Psoriasis Area Severity Index (PASI) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease).
Part 1 and Part 2: Change from Baseline in Absolute Psoriasis Area and Severity Index (PASI) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Absolute Body Surface Area (BSA) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%).
Part 1 and Part 2: Change from Baseline in Absolute Body Surface Area (BSA) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%). Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Percentage of Participants Achieving Physician Global Assessment (PGA) Score of 0 or 1 | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The PGA score is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score.
Part 1 and Part 2: Percentage of Participants Achieving Scalp Physician Global Assessment (scPGA) Score of 0 or 1 | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The scPGA score is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed.
Part 1 and Part 2: Percentage of Participants Achieving Palmoplantar Physician's Global Assessment (PPPGA) Score of 0 or 1 | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The PPPGA score is used to assess the average severity of psoriasis lesions on hands and/or feet. The PPPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe psoriasis lesions on hands and/or feet. Only in participants with palmar or plantar involvement the PPPGA assessment will be performed.
Part 1 and Part 2: Absolute Physician Global Assessment (PGA) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The PGA score is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score.
Part 1 and Part 2: Absolute Scalp Physician Global Assessment (scPGA) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The scPGA score is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed.
Part 1 and Part 2: Absolute Palmoplantar Physician's Global Assessment (PPPGA) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The PPPGA score is used to assess the average severity of severity of psoriasis lesions on hands and/or feet. The PPPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe psoriasis lesions on hands and/or feet. Only in participants with palmar or plantar involvement the PPPGA assessment will be performed.
Part 1 and Part 2: Change from Baseline in Absolute Physician Global Assessment (PGA) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The PGA score is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Change from Baseline in Absolute Scalp Physician Global Assessment (scPGA) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The scPGA score is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Change from Baseline in Absolute Palmoplantar Physician's Global Assessment (PPPGA) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The PPPGA score is used to assess the average severity of psoriasis lesions on hands and/or feet. The PPPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe psoriasis lesions on hands and/or feet. Only in participants with palmar or plantar involvement the PPPGA assessment will be performed. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Percentage of Participants Achieving Dermatology Quality of Life Index (DLQI) Score of 0 or 1 | Part 1: Weeks 8 and 16; Part 2: Weeks 32 and 40
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Part 1 and Part 2: Absolute Dermatology Quality of Life Index (DLQI) Score | Part 1: Weeks 8 and 16; Part 2: Weeks 32 and 40
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Part 1 and Part 2: Change from Baseline in Absolute Dermatology Quality of Life Index (DLQI) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: Baseline, Weeks 32 and 40
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Absolute Skindex-16 Score | Part 1: Weeks 8 and 16; Part 2: Weeks 32 and 40
  Skindex is the dermatological instruments to measure dermatology-specific Health-Related Quality of Life (HRQoL). The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1-4), emotions (5-11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (never bothered) to 6 (always bothered) with a total possible score ranging from 0 (best HRQoL) to 96 (worst HRQoL). Each item is then transformed to a linear scale from 0 to 100.
Part 1 and Part 2: Change from Baseline in Absolute Skindex-16 Score | Part 1: Baseline, Weeks 8 and 16; Part 2: Baseline, Weeks 32 and 40
  Skindex is the best dermatological instruments to measure dermatology-specific Health-Related Quality of Life (HRQoL). The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1-4), emotions (5-11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (never bothered) to 6 (always bothered) with a total possible score ranging from 0 (best HRQoL) to 96 (worst HRQoL). Each item is then transformed to a linear scale from 0 to 100. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Absolute Pruritus-Visual Analogue Scale (VAS) Score | Part 1: Weeks 8 and 16; Part 2: DMF: Weeks 24, 36 and 40, Tildrakizumab: Weeks 20, 32 and 40
  The pruritus-VAS is used to assess the pruritus by ticking the scale, which describes pruritus the best. The pruritus-VAS is a single-item continuous scale comprised of a 10 centimeter (cm) [(100 millimeter (mm)] horizontal/vertical line anchored by two verbal descriptors, one for each symptom extreme. For pruritus intensity, the scale is anchored by "no pruritus" (score of 0) and "worst imaginable pruritus" (score of 100 mm).
Part 1 and Part 2: Change from Baseline in Absolute Pruritus-Visual Analogue Scale (VAS) Score | Part 1: Baseline, Weeks 8 and 16; Part 2: Baseline, DMF: Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The pruritus-VAS is used to assess the pruritus by ticking the scale, which describes pruritus the best. The pruritus-VAS is a single-item continuous scale comprised of a 10 centimeter (cm) [(100 millimeter (mm)] horizontal/vertical line anchored by two verbal descriptors, one for each symptom extreme. For pruritus intensity, the scale is anchored by "no pruritus" (score of 0) and "worst imaginable pruritus" (score of 100 mm). Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 1 and Part 2: Absolute Medical Outcomes Study (MOS) Score | Part 1: Week 16; Part 2: Week 40
  The MOS score questionnaire consists of 12 items leading to 6 subscales or domains: sleep disturbance, sleep adequacy, daytime sleepiness, 'supposed or known' snoring, being awakened by shortness of breath or by a headache, and quantity of sleep. Subscales are standardised to yield scores from 0 to 100, with the exception of sleep quantity. Higher scores on the MOS score reflects more of the attribute indicated by the subscale name.
Part 1 and Part 2: Change from Baseline in Absolute Medical Outcomes Study (MOS) Score | Part 1: Baseline, Week 16; Part 2: Baseline, Week 40
  The MOS score questionnaire consists of 12 items leading to 6 subscales or domains: sleep disturbance, sleep adequacy, daytime sleepiness, 'supposed or known' snoring, being awakened by shortness of breath or by a headache, and quantity of sleep. Subscales are standardised to yield scores from 0 to 100, with the exception of sleep quantity. Higher scores on the MOS score reflects more of the attribute indicated by the subscale name. Baseline value is defined as values collected at Week 1 of Part 1 of the study. Change from baseline will be calculated by subtracting post-dose value baseline value.
Part 2: Percent Change from Baseline in Absolute Psoriasis Area Severity Index (PASI) Score | DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Physician Global Assessment (PGA) Score | DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  PGA is used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Scalp Physician Global Assessment (scPGA) Score | DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The scPGA scores is used to assess the average severity of scalp psoriasis lesions. The scPGA is also 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe scalp psoriasis lesions. Only in participants with scalp involvement, the scPGA assessment will be performed. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Palmoplantar Physician's Global Assessment (PPPGA) Score | DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  PPPGA Scores is used to assess the average severity of psoriasis lesions on hands and/or feet. The PPPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), where higher score indicates severe psoriasis lesions on hands and/or feet. Only in participants with palmar or plantar involvement the PPPGA assessment will be performed. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Dermatology Quality of Life Index (DLQI) Score | Baseline, Weeks 32 and 40
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Skindex-16 Score | Baseline, Weeks 32 and 40
  Skindex is the dermatological instruments to measure dermatology-specific Health-Related Quality of Life (HRQoL). The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1-4), emotions (5-11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (never bothered) to 6 (always bothered) with a total possible score ranging from 0 (best HRQoL) to 96 (worst HRQoL). Each item is then transformed to a linear scale from 0 to 100. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Pruritus-Visual Analogue Scale (VAS) Score | DMF: Baseline, Weeks 24, 36 and 40, Tildrakizumab: Baseline, Weeks 20, 32 and 40
  The pruritus-VAS is used to assess the pruritus by ticking the scale, which describes pruritus the best. The pruritus-VAS is a single-item continuous scale comprised of a 10 centimeter (cm) [(100 millimeter (mm)] horizontal/vertical line anchored by two verbal descriptors, one for each symptom extreme. For pruritus intensity, the scale is anchored by "no pruritus" (score of 0) and "worst imaginable pruritus" (score of 100 mm). Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Percent Change from Baseline in Absolute Medical Outcomes Study (MOS) Score | Baseline, Week 40
  The MOS score questionnaire consists of 12 items leading to 6 subscales or domains: sleep disturbance, sleep adequacy, daytime sleepiness, 'supposed or known' snoring, being awakened by shortness of breath or by a headache, and quantity of sleep. Subscales are standardised to yield scores from 0 to 100, with the exception of sleep quantity. Higher scores on the MOS score reflects more of the attribute indicated by the subscale name. Baseline value is defined as values collected at Week 1 of Part 1 of the study.
Part 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From start of study drug administration up to Week 49
  An Adverse event (AE) is defined as "any untoward medical occurrence in a clinical trial participant (regardless of the administration of the study drug and its causal relationship to it). An AE can therefore be any unfavourable and unintended medical occurrence during the participant's participation in the trial, including deterioration of a pre-existing medical condition, an abnormal clinically significant finding in a laboratory assessment, or an abnormal clinically significant finding in the physical examination or vital sign. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward will be counted as TEAE.
Percentage of Participants Withdrawing from Trial | From start of study drug administration up to Week 49
Number of Participants with Treatment Compliance | From start of study drug administration up to Week 49
Percentage of Participants Using Topical Corticosteroids (TCS) | Part 1: Baseline up to Week 14; Part 2: Week 20 to Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, SAS
Locations (3):
- Investigator Site 3, Augsburg, Germany
- United Kingdom (2):
  - Investigator Site 1, Bristol
  - Investigator Site 2, London